CLINICAL TRIAL: NCT00159614
Title: Effect of KW-3902IV in Combination With IV Furosemide on Renal Function in Subjects With Congestive Heart Failure (CHF) and Renal Impairment
Brief Title: Effect of KW-3902IV in Combination With IV Furosemide on Renal Function in Subjects With CHF and Renal Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NovaCardia, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CKI-203
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Heart Failure, Congestive; Renal Insufficiency
Keywords: renal insufficiency; diuretic; heart failure, congestive
MeSH Terms: conditions — Heart Failure; Renal Insufficiency

INTERVENTIONS:
Drug: KW-3902IV

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of KW-3902IV and measure its effect on renal function.

ELIGIBILITY:
Inclusion Criteria:

* Stable congestive heart failure
* Impaired renal function
* Taking oral loop diuretic

Exclusion Criteria:

* Acutely decompensated (unstable) and end stage heart failure
* Diuretics other than loop diuretics
* Pregnant or nursing
* Inability to follow instructions
* Participation in another clinical trial within past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-09

PRIMARY OUTCOMES:
Comparison of KW-3902IV alone or with loop diuretic on renal function.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - San Diego, California
  - Baltimore, Maryland
  - Ayer, Massachusetts
  - Boston, Massachusetts
  - Kalamazoo, Michigan
  - Tullahoma, Tennessee

REFERENCES:
- [Derived] Dittrich HC, Gupta DK, Hack TC, Dowling T, Callahan J, Thomson S. The effect of KW-3902, an adenosine A1 receptor antagonist, on renal function and renal plasma flow in ambulatory patients with heart failure and renal impairment. J Card Fail. 2007 Oct;13(8):609-17. doi: 10.1016/j.cardfail.2007.08.006. PMID 17923351